CLINICAL TRIAL: NCT00611702
Title: Genomics of Chronic Renal Allograft Rejection
Brief Title: Genomics of Chronic Renal Allograft Rejection (The GoCAR Study)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT GTCRP-01
Record Dates: First submitted 2008-02-07; First posted 2008-02-11 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Transplantation
Keywords: ELISPOT; RT-PCR; Luminex; Genomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood from both kidney donor and recipient and transplant kidney biopsy samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Kidney biopsy — Kidney biopsy (recipients only) will be obtained for RT-PCR, microarray analyses and histology.

SUMMARY:
Doctors have had success preventing certain types of kidney transplant rejection by suppressing the immune system. However, an individual's genetic make-up and the strength of an immune response to a transplant may also determine whether a transplanted organ is rejected. The purpose of this study is to look at the genetic profile and immune response of people who have had kidney transplants and to correlate the findings with kidney transplant rejection episodes. Donor genetic profiles will also be studied and correlated with the recipient's information.

DETAILED DESCRIPTION:
New immunosuppressive drugs have improved short-term transplant survival but have not affected long-term transplant survival. Rejection is caused by both immunological and non-immunological factors from both the donor and the recipient. Although the exact cause of chronic rejection is not known, it is associated with the presence of C4d, a degradation product of the antibody response cascade, and the presence of circulating donor-specific antibodies (DSAs). The purpose of this study is to determine the role of cell- and antibody-mediated responses in chronic rejection of transplants, to determine the gene expression profile associated with the development of chronic rejection, and to determine whether variants of specific genes cause susceptibility to rejection.

This is an observational study of people who will be receiving kidney transplants and participants will be followed for 2 years. Study visits for kidney transplant recipients will occur at study entry and at months 3, 6, 12, 18, and 24 after transplant. At these visits, adverse event assessment, rejection assessment, medication history questionnaire, and blood collection will occur. At some visits, a physical exam and a kidney biopsy will occur. Blood will also be collected from living kidney donors at the time of donation if both donor and recipient agree to be in the study. This study will be take place at 4 clinical sites: Mount Sinai School of Medicine, University of Wisconsin-Madison, Westmead Hospital, and Northwestern Memorial Hospital. Brigham and Women's Hospital and Massachusetts General Hospital will also participate in the study as central laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidates from living or deceased donors
* Male or female, ages 18-75 years
* Subject must be able to understand and provide written informed consent
* Living Donors - Recipient also consents to participate in the study

Exclusion Criteria:

* Presence of Donor Specific Antibodies in living donor recipients prior to transplantation OR positive cross match according to site-specific technique in cadaveric donor recipients
* Recipients of multiple organ transplants, with the exception of kidney/pancreas transplants.
* Inability or unwillingness to comply with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals receiving a kidney transplant and individuals who are donating a kidney
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2008-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Correlation of chronic rejection with patterns and intensity of recipient alloreactivity | Throughout study
Correlation of chronic rejection with recipient gene expression profiles | Throughout study
Correlation of chronic rejection with polymorphic variants of specific susceptibility genes in donor and recipient | Throughout study

SECONDARY OUTCOMES:
Correlation of the development of donor specific antibodies after transplant and/or the presence of C4d staining with patterns and intensity of recipient alloreactivity | Throughout study
Correlation of the development of donor specific antibodies after transplant and/or the presence of C4d staining with recipient gene expression profiles | Throughout study
Correlation of the development of donor-specific antibodies after transplant and/or the presence of C4d staining of peritubular basement membranes on renal biopsy with polymorphic variants of specific susceptibility genes in donor and recipient | Throughout study
Correlation of the development of donor-specific antibodies after transplant and/or the presence of C4d staining of peritubular basement membranes on renal biopsy with chronic rejection | Throughout study
Correlation of the development of donor-specific antibodies after transplant and/or the presence of C4d staining of peritubular basement membranes on renal biopsy allograft dysfunction as defined by the protocol | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Barbara T. Murphy, MD, Principal Investigator — Division of Nephrology, Mt. Sinai School of Medicine
Locations (5):
- United States (4):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Mt. Sinai School of Medicine, New York, New York
  - University of Wisconsin-Madison, Madison, Wisconsin
- Westmead Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Vitalone MJ, O'Connell PJ, Wavamunno M, Fung CL, Chapman JR, Nankivell BJ. Transcriptome changes of chronic tubulointerstitial damage in early kidney transplantation. Transplantation. 2010 Mar 15;89(5):537-47. doi: 10.1097/TP.0b013e3181ca7389. PMID 20147884
- [Background] Vitalone MJ, O'Connell PJ, Jimenez-Vera E, Yuksel A, Wavamunno M, Fung CL, Chapman JR, Nankivell BJ. Epithelial-to-mesenchymal transition in early transplant tubulointerstitial damage. J Am Soc Nephrol. 2008 Aug;19(8):1571-83. doi: 10.1681/ASN.2007050580. Epub 2008 May 14. PMID 18480317
- [Background] Dinavahi R, George A, Tretin A, Akalin E, Ames S, Bromberg JS, Deboccardo G, Dipaola N, Lerner SM, Mehrotra A, Murphy BT, Nadasdy T, Paz-Artal E, Salomon DR, Schroppel B, Sehgal V, Sachidanandam R, Heeger PS. Antibodies reactive to non-HLA antigens in transplant glomerulopathy. J Am Soc Nephrol. 2011 Jun;22(6):1168-78. doi: 10.1681/ASN.2010111183. Epub 2011 May 12. PMID 21566057
- [Background] Kruger B, Krick S, Dhillon N, Lerner SM, Ames S, Bromberg JS, Lin M, Walsh L, Vella J, Fischereder M, Kramer BK, Colvin RB, Heeger PS, Murphy BT, Schroppel B. Donor Toll-like receptor 4 contributes to ischemia and reperfusion injury following human kidney transplantation. Proc Natl Acad Sci U S A. 2009 Mar 3;106(9):3390-5. doi: 10.1073/pnas.0810169106. Epub 2009 Feb 13. PMID 19218437
- [Background] Wavamunno MD, O'Connell PJ, Vitalone M, Fung CL, Allen RD, Chapman JR, Nankivell BJ. Transplant glomerulopathy: ultrastructural abnormalities occur early in longitudinal analysis of protocol biopsies. Am J Transplant. 2007 Dec;7(12):2757-68. doi: 10.1111/j.1600-6143.2007.01995.x. Epub 2007 Oct 6. PMID 17924997
- [Background] Gurkan S, Luan Y, Dhillon N, Allam SR, Montague T, Bromberg JS, Ames S, Lerner S, Ebcioglu Z, Nair V, Dinavahi R, Sehgal V, Heeger P, Schroppel B, Murphy B. Immune reconstitution following rabbit antithymocyte globulin. Am J Transplant. 2010 Sep;10(9):2132-2141. doi: 10.1111/j.1600-6143.2010.03210.x. PMID 20883548
- [Background] Farris AB, Adams CD, Brousaides N, Della Pelle PA, Collins AB, Moradi E, Smith RN, Grimm PC, Colvin RB. Morphometric and visual evaluation of fibrosis in renal biopsies. J Am Soc Nephrol. 2011 Jan;22(1):176-86. doi: 10.1681/ASN.2009091005. Epub 2010 Nov 29. PMID 21115619
- [Background] Schroppel B, Kruger B, Walsh L, Yeung M, Harris S, Garrison K, Himmelfarb J, Lerner SM, Bromberg JS, Zhang PL, Bonventre JV, Wang Z, Farris AB, Colvin RB, Murphy BT, Vella JP. Tubular expression of KIM-1 does not predict delayed function after transplantation. J Am Soc Nephrol. 2010 Mar;21(3):536-42. doi: 10.1681/ASN.2009040390. Epub 2009 Dec 17. PMID 20019169
- [Background] Luan Y, Mosheir E, Menon MC, Wilson D, Woytovich C, Ochando J, Murphy B. Monocytic myeloid-derived suppressor cells accumulate in renal transplant patients and mediate CD4(+) Foxp3(+) Treg expansion. Am J Transplant. 2013 Dec;13(12):3123-31. doi: 10.1111/ajt.12461. Epub 2013 Sep 18. PMID 24103111
- [Derived] O'Connell PJ, Zhang W, Menon MC, Yi Z, Schroppel B, Gallon L, Luan Y, Rosales IA, Ge Y, Losic B, Xi C, Woytovich C, Keung KL, Wei C, Greene I, Overbey J, Bagiella E, Najafian N, Samaniego M, Djamali A, Alexander SI, Nankivell BJ, Chapman JR, Smith RN, Colvin R, Murphy B. Biopsy transcriptome expression profiling to identify kidney transplants at risk of chronic injury: a multicentre, prospective study. Lancet. 2016 Sep 3;388(10048):983-93. doi: 10.1016/S0140-6736(16)30826-1. Epub 2016 Jul 22. PMID 27452608
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/